CLINICAL TRIAL: NCT00580957
Title: The Autonomic Nervous System and the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 060085; CRC-1522 (Other: Vanderbilt University)
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
Keywords: Obesity; Hypertension; Autonomic Nervous System
MeSH Terms: conditions — Obesity; Hypertension | interventions — Dental Occlusion; Trimethaphan; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blocked (Experimental): Active treatment arm. Transient autonomic blockade with Trimethaphan and blood pressure restoration with L-NMMA will be used during insulin clamp
  Interventions: Drug: Blocked
- Intact (Placebo Comparator): Saline will be used instead of trimethaphan during insulin clamp
  Interventions: Drug: Intact

INTERVENTIONS:
Drug: Blocked — Trimethaphan 4 mg/min IV will be infused for the duration of the study. L-NMMA 125-500 mcg/k/min IV will be titrated to restore blood pressure to pre-trimethaphan levels Insulin clamp will be used to determine insulin resistance
  Other Names: Trimethaphan
  Arms: Blocked
Drug: Intact — Saline IV infusion to simulate trimethaphan infusion in active arm Insulin clamp will be done to determine insulin resistance
  Other Names: Saline
  Arms: Intact

SUMMARY:
The overall goal of this proposal is to determine the role of the autonomic nervous system in the insulin resistant state associated with obesity and the metabolic syndrome. Obesity results from an accumulation of excessive fat deposit due to increase caloric intake or decrease energy expenditure, this condition is usually associated with diseases such as hypertension or diabetes, a cluster known as the metabolic syndrome. The first step in the development of the metabolic syndrome is a resistance to the action of insulin. The mechanism underlying insulin resistance in obesity is still unknown, however some investigators have proposed that the autonomic nervous system, particularly the increase sympathetic activation in obesity may play an important role. We have extensive experience studying the role of the autonomic nervous system in the cardiovascular alterations associated with obesity by producing complete autonomic withdrawal with a drug named trimethaphan. We propose to use the same approach to study the role of the autonomic nervous system in the development of insulin resistance in obesity.

DETAILED DESCRIPTION:
The purpose of this study is to look at the role of the autonomic nervous system, an involuntary nervous system that controls your blood pressure, in insulin resistance and the metabolic syndrome. Insulin is a substance that helps your body use the sugar in the food that you eat. Some people's tissues stop reacting in a normal way to insulin, a condition known as insulin resistance. A person with insulin resistance can have other health problems, such as obesity, high cholesterol, and high blood pressure. These problems together are called the metabolic syndrome. We think that the autonomic or involuntary nervous system controls the way your body responds to insulin. This system is changed in obese people, and we think that it may cause the insulin resistance. We plan to study this with two drugs -trimethaphan and L-NMMA. Neither of these drugs are approved by the Food and Drug Administration (FDA), and they will be used for research purposes only.

Fifty people will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* For lean subjects:
* 21 subjects aged 18-60 yr.
* All potential volunteers will have routine blood test to screen for hepatic, renal, and hematological abnormalities.
* Body mass index < 25Kg/m^2 .
* Female volunteers of childbearing potential will undergo HCG pregnancy test at screening and again on the study day.
* For Obese subjects with metabolic syndrome:
* 21 subjects aged 18-60 yr.
* All potential volunteers will have routine blood test to screen for hepatic, renal, and hematological abnormalities.
* Body mass index > 30Kg/m^2.
* Participants will be enrolled if they met at least three of the following criteria for metabolic syndrome (Expert panel, Jama 2001):

  1. Waist circumference >102 cm in men and >88 cm in women
  2. High fasting blood sugar (>110 mg%)
  3. Triglyceride levels >150 mg%
  4. Low HDL cholesterol (<40 mg% for men; <50 mg% for women)
  5. High blood pressure (systolic=130 and diastolic = 85 mmHg) • Female volunteers of childbearing potential will undergo serum HCG pregnancy test at screening and urine HCG pregnancy test again on the study day.

Exclusion Criteria:

* Pregnant females
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs or anemic (anemia defined as Hcto less than 35%)
* Subjects with a recent medical illness documented by physicians's visit or detected during the screening visit.
* Subjects with a history of coronary heart disease.
* Subjects with known kidney or liver disease.
* Subjects with recent weight loss or consuming low carbohydrate diet.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Blocked: Active treatment arm. Transient autonomic blockade with Trimethaphan and blood pressure restoration with L-NMMA will be used during insulin clamp
  Blocked: Trimethaphan 4 mg/min IV will be infused for the duration of the study.
  L-NMMA 125-500 mcg/k/min IV will be titrated to restore blood pressure to pre-trimethaphan levels Insulin clamp will be used to determine insulin resistance
Period: Overall Study
Arm/Group | Blocked | Intact
Started | 28 | 28
Completed | 21 | 21
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Blocked Then Intact: Active treatment arm. Transient autonomic blockade with Trimethaphan and blood pressure restoration with L-NMMA will be used during insulin clamp
  Blocked: Trimethaphan 4 mg/min IV will be infused for the duration of the study.
  L-NMMA 125-500 mcg/k/min IV will be titrated to restore blood pressure to pre-trimethaphan levels Insulin clamp will be used to determine insulin resistance
- Intact Then Blocked: Saline will be used instead of trimethaphan during insulin clamp
  Intact: Saline IV infusion to simulate trimethaphan infusion in active arm Insulin clamp will be done to determine insulin resistance
- Total: Total of all reporting groups
Arm/Group | Blocked Then Intact | Intact Then Blocked | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (6) | 43 (5) | 43 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Insulin Resistance
Description: Glucose infusion rate in mg/kg/min
Time Frame: Last 30 minutes of a two hour insulin clamp
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Blocked | Intact
Number analyzed (Participants) | 21 | 21
mg/kg/min | 3.8 (0.3) | 3.1 (0.3)

ADVERSE EVENTS:
Time Frame: During and up to 1 hour after finishing the 2 hour insulin clamp.
Arm/Group | Blocked | Intact
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No